CLINICAL TRIAL: NCT07250880
Title: Evaluation of Serum Ceramides C16, C24, and Sphingosine-1-Phosphate (S1P) in Patients With Acne Vulgaris
Acronym: CER-S1P-ACNE
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dalia Ahmed Helmy Ahmed, Dermatology Resident At Albalyna central hospital, Sohag University
Other Study IDs: Soh-Med-25-10-11MS
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — sphingosine 1-phosphate; membrane-bound transcription factor peptidase, site 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples collected from venous blood. Samples will be processed by centrifugation and stored at -80°C until analysis. No DNA will be extracted from the specimens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Acne vulgaris patients: Both males and females aged 15-40 years.
  • Mild, Moderate, severe and very severe cases will be included
  Interventions: Other: Blood sample collection for biochemical analysis of serum ceramides (C16, C24) and sphingosine-1-phosphate (S1P).
- Healthy controls: Healthy controls
  Description:
  Age- and sex-matched healthy volunteers
  Interventions: Other: Blood sample collection for biochemical analysis of serum ceramides (C16, C24) and sphingosine-1-phosphate (S1P).

INTERVENTIONS:
Other: Blood sample collection for biochemical analysis of serum ceramides (C16, C24) and sphingosine-1-phosphate (S1P). — Venous blood samples (5 mL) will be collected from all participants under aseptic conditions. Serum will be separated and stored at -80°C until analysis. Quantitative estimation of ceramide C16, ceramide C24, and sphingosine-1-phosphate (S1P) will be performed using liquid chromatography-tandem mass spectrometry (LC-MS/MS). No therapeutic intervention will be given.

SUMMARY:
Acne vulgaris is a common chronic inflammatory skin disorder that affects adolescents and young adults. Recent research has shown that lipid mediators, including ceramides and sphingolipids, play an important role in maintaining skin barrier function and inflammation.

This study aims to evaluate the serum levels of ceramide C16, ceramide C24, and sphingosine-1-phosphate (S1P) in patients with acne vulgaris and compare them to healthy controls. The goal is to explore their possible role in the pathogenesis and severity of acne. Blood samples will be collected from participants, and quantitative analysis will be performed using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

DETAILED DESCRIPTION:
Acne vulgaris involves complex biochemical and immunologic mechanisms that extend beyond the traditional concepts of follicular obstruction and increased sebum production. Emerging evidence highlights the contribution of systemic lipid mediators-particularly sphingolipids-in influencing keratinocyte behavior, sebaceous gland activity, and inflammatory signaling pathways. Disturbances in circulating ceramides and their downstream metabolites may reflect dysregulated lipid homeostasis that parallels the clinical manifestations of acne.

In this study, specific attention is given to three sphingolipid biomarkers that have been increasingly linked to cutaneous biology: Ceramide C16, Ceramide C24, and Sphingosine-1-phosphate (S1P). These molecules participate in cell differentiation, apoptosis, and immune responses, and their altered levels may provide insight into acne-related metabolic shifts. By quantitatively assessing their serum concentrations in affected individuals and comparing them with healthy subjects, the study aims to characterize potential biochemical patterns associated with disease presence and activity.

All biological samples will be processed using a validated LC-MS/MS analytical platform to ensure precise measurement of each sphingolipid species. The findings may help to clarify whether systemic sphingolipid disturbances contribute to acne pathophysiology and could support the development of lipid-based biomarkers or therapeutic strategies in future dermatologic research.

ELIGIBILITY:
Inclusion Criteria:

* For Case Group

This group will consist of (40) patients :

* Both males and females aged 15-40 years.
* Mild, Moderate, severe and very severe cases will be included. 5

For Control Group:

• This group will consist of age- and sex-matched (40) healthy volunteers.

Exclusion Criteria:

* Presence of any dermatological condition other than acne vulgaris (for cases).

  * Use of systemic or topical treatment such as isotretinoin or antibiotics within the last 3 months.
  * Pregnancy or lactation.
  * History of lipid-lowering therapy or supplements affecting ceramide or sphingolipid metabolism.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study Population:
  A. Inclusion Criteria:
  For Case Group
  This group will consist of (40) patients :
  * Both males and females aged 15-40 years.
  * Mild, Moderate, severe and very severe cases will be included. 5
  For Control Group:
  • This group will consist of age- and sex-matched (40) healthy volunteers.
  B. Exclusion Criteria (for both groups):
  * Presence of any dermatological condition other than acne vulgaris (for cases).
  * Use of systemic or topical treatment such as isotretinoin or antibiotics within the last 3 months.
  * Pregnancy or lactation.
  * History of lipid-lowering therapy or supplements affecting ceramide or sphingolipid metabolism
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Serum levels of Ceramide C16, Ceramide C24, and Sphingosine-1-Phosphate (S1P) | At baseline (single visit)
  Quantitative assessment of serum concentrations of Ceramide C16, Ceramide C24, and Sphingosine-1-Phosphate (S1P) in acne vulgaris patients and healthy controls using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

DOCUMENTS (1):
  • Study Protocol (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT07250880/Prot_000.pdf